CLINICAL TRIAL: NCT00062803
Title: The Van Gogh-PE Trial, a Multicenter, International, Randomized, Open-Label, Assessor-Blind, Non-Inferiority Study Comparing the Efficacy and Safety of Once-Weekly Subcutaneous SR34006 With the Combination of (LMW)Heparin and Vitamin K Antagonist (VKA) in the Treatment of Acute Symptomatic Pulmonary Embolism
Brief Title: SR34006 Compared to Vitamin K Antagonist (VKA) in the Treatment of Pulmonary Embolism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EFC3484
Record Dates: First submitted 2003-06-16; First posted 2003-06-17 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — idraparinux; Dalteparin

INTERVENTIONS:
Drug: SR34006
Drug: (LMW)heparin
Drug: Warfarin VKA
Drug: Acenocoumarol VKA

SUMMARY:
Patients who have a pulmonary embolism (blood clot in the lung) will be treated in this study. The purpose of the study is to compare the safety and effectiveness of a new injectable anticoagulant (blood-thinning) drug, SR34006, with the standard way of treating a pulmonary embolism. The standard treatment includes injections or infusions of an anticoagulant drug, (LMW)heparin, for about a week followed by anticoagulant tablets (warfarin or acenocoumarol) which are taken by mouth.

Assignment to either SR34006 or (LMW)heparin plus warfarin or acenocoumarol will be purely by chance and will be known by both patients and their doctors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute symptomatic Pulmonary Embolism (PE) with or without concomitant Deep Vein Thrombosis (DVT)
* Written informed consent

Exclusion Criteria:

* Legal lower age limitations (country specific)
* Thrombectomy, insertion of a caval filter, or use of a fibrinolytic agent to treat the current episode of PE
* Other indication for VKA than PE/DVT
* More than 36 hours pre-randomization treatment with therapeutic dosages of (LMW)heparin or initiation of VKA treatment prior to randomization
* Participation in another pharmacotherapeutic study within the prior 30 days
* Creatinine clearance <10 mL/min, severe hepatic disease, or bacterial endocarditis
* Life expectancy <3 months
* Active bleeding or high risk for bleeding
* Uncontrolled hypertension: systolic blood pressure >180 mm Hg or diastolic blood pressure >110 mm Hg
* Pregnancy or childbearing potential without proper contraceptive measures or women who are breastfeeding
* Any other contraindication listed in the labeling of warfarin, acenocoumarol, unfractionated heparin, enoxaparin, or tinzaparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
symptomatic recurrent pulmonary embolism or deep vein thrombosis within 3 months.

SECONDARY OUTCOMES:
symptomatic recurrent PE/DVT within 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (93):
- United States (54):
  - Jerry L. Pettic VA Medical Center, Loma Linda, California
  - University of California, San Diego Medical Center, San Diego, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Colorado Hospital, Denver, Colorado
  - Bay Pines VA Medical Center, Bay Pines, Florida
  - Brandon Regional Hospital, Brandon, Florida
  - Holmes Regional Medical Center, Melbourne, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - St. Joseph's Hospital, Tampa, Florida
  - Medical College of Georgia, Augusta, Georgia
  - DeKalb Medical Center, Decatur, Georgia
  - Loyola University Medical Center and Outpatient Clinic, Maywood, Illinois
  - Olathe Medical Center, Olathe, Kansas
  - Christus St. Patrick Hospital, Lake Charles, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - St. Joseph Mercy - Oakland, Pontiac, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Lovelace Health Systems, Clinical Thrombosis Center, Albuquerque, New Mexico
  - Winthrop Pulmonary Associates, Mineola, New York
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai School of Medicine, New York, New York
  - St. Luke's-Roosevelt Hospital Center, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Altru Health System Hospital, Grand Forks, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Medical College of Ohio, Toledo, Ohio
  - Saint Anthony Hospital, Oklahoma City, Oklahoma
  - Oklahoma City VA Medical Center, Oklahoma City, Oklahoma
  - OU Medical Center, Oklahoma City, Oklahoma
  - INTEGRIS Southwest Medical Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Crozer-Chester Medical Center, Upland, Pennsylvania
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Mary Black Memorial Hospital, Spartanburg, South Carolina
  - Baptist Memorial Hospital Memphis, Memphis, Tennessee
  - The West Cancer Clinic, Memphis, Tennessee
  - Northwest Texas Healthcare System, Amarillo, Texas
  - The Methodist Hospital, Houston, Texas
  - Scott & White Memorial Hospital & Clinic, Temple, Texas
  - The University of Texas Health Center at Tyler, Tyler, Texas
  - University Hospital, Salt Lake City, Utah
  - Inova Alexandria Hospital, Alexandria, Virginia
  - MedSource, Inc., Chesapeake, Virginia
  - Portsmouth Pulmonary Associates, Chesapeake, Virginia
  - Pulmonary Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - Maryview Medical Center, Portsmouth, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Sacred Heart Medical Center, Spokane, Washington
- Buenos Aires, Argentina
- Australia (2):
  - Box Hill, Clayton, Garran, Kogarah, Ringwood East
  - Saint Leonards, South Australia
- Graz, Austria
- Bruxelles, Charleroi, Leuven, Liege, Yvoir, Belgium
- Goiania, Porto Alegre, Sao Paulo, Salvador, Brazil
- Canada (12):
  - University of Alberta Hospital, Edmonton, Alberta
  - Kelowna General Hospital, Kelowna, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - Hamilton Health Sciences - General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - University Health Network, Toronto General Hospital, Toronto, Ontario
  - Humber River Regional Hospital, Weston, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Hotel-Dieu de St-Jerome, Saint-Jérôme, Quebec
- Czechia (2):
  - Brno, Jihlava, Karlovy Vary, Kladno, Ostrava Poruba, Prague
  - Pilsen
- Denmark (2):
  - Arhus, Frederiksberg, Glostrup, Hillerod, Kobenhavn, Odense
  - Roskilde
- Hus, Jyvaskyla, Seinajoki, Turku, Finland
- France (4):
  - Armentieres, Besancon, Bethune, Brest, Chambray Les Tours
  - Clamart, Lens, Lille, Nice, Nimes, Paris, Rennes, Roubaix
  - Saint Malo, Valenciennes
  - Tourcoing
- Germany (2):
  - Augsburg, Berlin, Bochum, Dresden, Garmisch-Partenkirchen
  - Heidelberg, Ibbenburen, Mannheim, Munchen
- Italy (2):
  - Cremona, Fidenza, Genova, Lecco, Milano, Padova, Parma, Pavia
  - Piacenza, Pisa, Reggio Emilia, Treviso, Venezia
- Netherlands (2):
  - Alkmaar, Amersfoort, Amsterdam, Breda, Gouda, Groningen
  - Haarlem, Maastricht, Nieuwegein
- Oslo, Rud, Norway
- Lublin, Warszawa, Wroclaw, Poland
- Badalona, Madrid, Sevilla, Spain
- Goteborg, Jonkoping, Stockholm, Varnamo, Sweden
- Basel, Bern, Lugano, Switzerland
- London, United Kingdom

REFERENCES:
- [Derived] Prins MH, Guillemin I, Gilet H, Gabriel S, Essers B, Raskob G, Kahn SR. Scoring and psychometric validation of the Perception of Anticoagulant Treatment Questionnaire (PACT-Q). Health Qual Life Outcomes. 2009 Apr 7;7:30. doi: 10.1186/1477-7525-7-30. PMID 19348685
- [Derived] van Gogh Investigators; Buller HR, Cohen AT, Davidson B, Decousus H, Gallus AS, Gent M, Pillion G, Piovella F, Prins MH, Raskob GE. Idraparinux versus standard therapy for venous thromboembolic disease. N Engl J Med. 2007 Sep 13;357(11):1094-104. doi: 10.1056/NEJMoa064247. PMID 17855670
- See also: Related Info — http://www.sanofi-aventis.com